CLINICAL TRIAL: NCT04210921
Title: Clinical Efficacy of Acupuncture in the Treatment of Temporomandibular Disorders(TMD)
Brief Title: Clinical Efficacy of Acupuncture in the Treatment of Temporomandibular Disorders (TMD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Li bin, Acupuncture director, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018BL-060-01
Record Dates: First submitted 2019-11-08; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Temporomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): In the treatment group, the Park needle with a real acupuncture will be penetrated in an appropriate angle into a depth of 10-15 mm. Acupuncture manually manipulated by lifting, thrusting, and twirling methods to produce a characteristic sensation known as "De Qi" (feeling of needle sensation refers to tenseness around the needle felt by the practitioner and numbness, distension, soreness, and heaviness around the point felt by the patient), and needles will be stimulated manually at least 10 s, then the needles will be retained for 30 minutes.
  Interventions: Device: Acupuncture
- Control group (Placebo Comparator): In the control group, the Park sham needle will instead of the real needle. It is retractile and adopts the sleeve type blunt needle design. When the blunt needle goes through the adhesive and contact with skin, it will move back into the hollow centre of the handle rather than penetrate into skin. The sham needle may be manipulated by lifting, thrusting or twirling as the real one, but it will not insert into the skin authentically.
  Interventions: Device: The park sham needle

INTERVENTIONS:
Device: Acupuncture — The acupuncture will be penetrated in an appropriate angle into a depth of 10-15 mm. Acupuncture manually manipulated by lifting, thrusting, and twirling methods to produce a characteristic sensation known as "De Qi" .
  Arms: Treatment group
Device: The park sham needle — When the blunt needle goes through the adhesive and contact with skin, it will move back into the hollow centre of the handle rather than penetrate into skin.
  Arms: Control group

SUMMARY:
This is a single-blinded, randomized controlled trial to explore the effectiveness of acupuncture in the treatment of the pain due to TMD using the latest diagnostic criteria combined with subjective and objective indexes.

DETAILED DESCRIPTION:
This is a single-blinded, randomized controlled clinical trial. A total of 60 participants will be randomly assigned to two different groups. The treatment group will receive acupuncture with real penetration of the needle, while participants in the control group will be treated with the Park sham needle. All participants will be given for 4 weeks of treatment and 4 weeks of follow-up.The primary end-point is the reducing in intensity of pain due to TMD, which will be evaluated before treatment, 4 weeks after treatment and follow-up (4 weeks after treatment) by using 0-10 visual analogue score. Secondary end points include Graded Chronic Pain Scale Version 2.0(GCPS 2.0),Jaw Functional Limitations Scale - 20-item (JFLS-20),Depression, Anxiety and Stress Scales (DASS-21),Pittsburgh sleep quality index (PSQI),Pressure Pain Threshold (PPT),Surface electromyogram(sEMG).

ELIGIBILITY:
Inclusion Criteria:

1. Pain disorders in accordance with Diagnostic Criteria for Temporomandibular Disorders (DC/TMD)
2. Pain in the jaw, temple, in the ear, in front of ear or headache in the temple at any sides, and pain or headache modified (remission or aggravation) with movement at least 3 months.
3. Cooperated in completing the clinical trial successfully without language and mental disorders.

Exclusion Criteria:

1. Conditions that result in regional pain in temporomandibular joint.
2. Autoimmune diseases that result in regional pain in the temporomandibular joint.
3. Mental illness or substance abuse.
4. Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale(VAS) | Baseline,Week- 4(treatment period) and Week-8(follow-up period)
  VAS is an international scale which reflects pain intensity and it has a 10-cm line ranging from 0 cm (no pain at all) to 10 cm (extremely painful). Pain intensity or pain relief in the tempormandibular joints will be measured by VAS. And then the investigators will compare the change of different time frames.The total score of this index is 10, and the better effect with the lower score.

SECONDARY OUTCOMES:
Graded Chronic Pain Scale Version 2.0(GCPS 2.0) | Baseline,Week- 4(treatment period) and Week-8(follow-up period)
  This scale includes the description of the degree of pain, a description of function, and a description of the time period of pain, which will provide effective data of the degree of pain within 1 month.The result of the index is divided into 5 grades. The less pain and influence with the lower the grade.
Jaw Functional Limitations Scale - 20-item (JFLS-20) | Baseline,Week- 4(treatment period) and Week-8(follow-up period)
  This scale includes the evaluation of mastication limitation, the evaluation of vertical mobility limitation, the evaluation of verbal and nonverbal communication limitation.There are 20 items in this index, with a total score of 200 points. The better the mandibular function with the lower the score.
Depression, Anxiety and Stress Scales (DASS-21) | Baseline,Week- 4(treatment period) and Week-8(follow-up period)
  This scale consists of three parts, 21 items in total. The total score of each part is 21 points. Less emotional distress with the lower the score.
Pittsburgh sleep quality index (PSQI) | Baseline,Week- 4(treatment period) and Week-8(follow-up period)
  The total score of this scale is 21. The better the sleep quality with the lower score.
Pressure Pain Threshold (PPT) | Baseline and Week- 4(treatment period)
  Participants will sit comfortably and relax their muscles during this measurement. A needle will be pressed at a constant speed perpendicular to the skin (0.5kg /cm2/second).The evaluator will be informed as soon as the participants feel pain and then record the results of measurement. The treatment is effective If the participants show elevated PPT after 4 weeks of treatment.
Surface electromyogram(sEMG) | Baseline and Week- 4(treatment period)
  The electrodes will be placed parallel to the muscle fibers of the specify what muschemuscle.EMG signal acquisition will be performed in three tasks: mandibular resting position (MR), during maximal voluntary contraction (MVC), and during habitual chewing (HC).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine affiliated to the Capital Medical University, Beijing, China